CLINICAL TRIAL: NCT04730271
Title: Comparison of Alignment Achieved Using the VELYS Robotic-Assisted Solution Versus Manual Instrumentation in Total Knee Arthroplasty: A Prospective, Non-Randomized Multi-Center Post-market Clinical Investigation
Brief Title: Comparison of Alignment Achieved Using the VELYS Robotic-Assisted Solution Versus Manual Instrumentation in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: DSJ_2019_08
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Osteo Arthritis Knee; Osteoarthritis
Keywords: Arthroplasty; Knee; Robotic-Assisted; VELYS; Accuracy
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Quantitative analysis of the X-rays will be conducted by a third party who will be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Manual Arm (Active Comparator): Subjects enrolled into this arm of the study will receive an ATTUNE primary total knee replacement that has been implanted using manual instrumentation which is the current standard of care at the participating sites.
  Interventions: Device: Total Knee Replacement
- Robotic-Assisted Arm (Experimental): Subjects enrolled into this arm will receive an ATTUNE primary total knee replacement that has been implanted with the use of the VELYS Robotic-Assisted Solution device.
  Interventions: Device: Total Knee Replacement

INTERVENTIONS:
Device: Total Knee Replacement — Subjects will be implanted with an ATTUNE Primary total knee replacement.

SUMMARY:
The purpose of this post-market research study is to gather clinical and radiographic (X-ray) information about total knee replacement surgeries completed with the VELYS Robotic-Assisted Solution and with standard manual instrumentation. The VELYS Robotic-Assisted Solution helps the surgeon to plan bone cuts and then accurately achieve the planned cuts during the total knee replacement surgery. The study aims to compare how well the VELYS Robotic-Assisted system enables the surgeon to position the implants exactly as planned compared to manual instrumentation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female and between the ages of 22 and 85 years at the time of consent, inclusive.
2. Subject has a severely painful and/or severely disabled joint resulting from osteoarthritis, post-traumatic arthritis or rheumatoid arthritis and in the opinion of the Investigator, is a suitable candidate for primary TKA using the devices described in this CIP with either resurfaced or non-resurfaced patellae.
3. Subject that is willing to give voluntary, written informed consent to participate in this clinical investigation and authorize the transfer of his/her information to the Sponsor
4. Subject is currently not permanently bedridden, as determined by the Investigator
5. Subject, in the opinion of the Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedures and follow-up visits and co-operate with investigational procedures.
6. Subject is able to read and comprehend the Informed Consent Document as well as complete the required PROs in English.
7. Subject's pre-operative alignment is such that (in the opinion of the Investigator) it is appropriate for it to be adjusted to mechanical long leg alignment during surgery.

Exclusion Criteria:

1. The Subject is a woman who is pregnant or lactating.
2. Contralateral knee has already been enrolled in this study.
3. Subject had a contralateral amputation.
4. Previous partial knee replacement (unicompartmental, bicompartamental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
5. Subject has an active local or systemic infection
6. Subject has loss of bone or musculature, osteoporosis, neuromuscular compromise or vascular deficiency in the affected limb in sufficient degree to render the procedure unjustifiable in the opinion of the Investigator (e.g. absence of musculo-ligamentous supporting structures, joint neuropathy)
7. Subject has severe instability secondary to advanced loss of osteochondral structure or the absence of collateral ligament integrity.
8. Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three (3) months.
9. Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Leslie, PhD, Study Director — DePuy Synthes
Locations (5):
- United States (5):
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Cuyuna Regional Medical Center, Crosby, Minnesota
  - OrthoCarolina, Charlotte, North Carolina
  - Campbell Clinic, Germantown, Tennessee
  - Proliance Orthopedic Associates, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 200 subjects were recruited into the study and received the intended treatment. An additional 34 subjects were recruited during the study but did not receive the planned treatment and were withdrawn and replaced in the study as allowed in the protocol.
Pre-assignment Details: Of the 34 subjects withdrawn without receiving the planned treatment, 8 were withdrawn due to a significant delay in having their procedure performed, 7 were withdrawn due to not meeting the inclusion/exclusion criteria, 6 were withdrawn due to the surgeon using an out of scope implant, 4 withdrew due to their insurance not covering surgery, 5 withdrew their consent, 3 were withdrawn due to the specified instrumentation not being available and one was withdrawn due to a change in the surgeon.
Groups:
- Study Arm: Robotic-Assisted
- Control Arm: Manual Instrumentation
Period: Overall Study
Arm/Group | Study Arm | Control Arm
Started (Enrolled and Treated) | 100 | 100
Intent to Treat and Completed 12 Week Follow up Per Protocol (Including required X-rays) | 90 | 92
Completed (Completed 1 year follow up (safety analysis set)) | 88 | 81
Not Completed | 12 | 19
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 7 | 13
Not completed — Lost to Follow-up | 3 | 3
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Knees
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm | Control Arm | Total
Number analyzed (Participants) | 100 | 100 | 200
Number analyzed (Knees) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (8.28) | 64.4 (9.05) | 65.5 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 53 | 101
  Male | 52 | 47 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 97 | 92 | 189
  Unknown or Not Reported | 0 | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 26 | 41
  White | 81 | 68 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of the Hip-Knee-Ankle Angle (HKA) Measured on Long-leg X-rays at 12 Weeks.
Description: The primary objective of this clinical investigation is to evaluate whether the accuracy to plan of the long leg alignment achieved with VELYS Robotic-Assisted Solution is non-inferior to the accuracy to plan of the long leg alignment achieved with the manual ATTUNE Intuition instrumentation. This will be assessed by measuring the Hip-Knee-Ankle angle (HKA) on long-leg X-rays taken at 12 weeks and comparing to the planned HKA. A smaller number represents improved accuracy and a better outcome.
Time Frame: 12 weeks
Population: Intent to Treat
Measure: Least Squares Mean (Standard Deviation); unit: Degrees
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 90 | 92
Degrees | 2.2 (1.77) | 2.5 (1.76)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; Test type: Non-Inferiority — Test of non-inferiority: Absolute value deviation from plan with ROBOTIC is less than it is with manual instruments (not using ROBOTIC) under a non-inferiority margin of 1.5 degrees; p < 0.0001, t-test, 1 sided

2. Secondary Outcome: Accuracy of the Distal Femoral Varus-valgus Angle Measured on Long Leg X-rays at 12 Weeks.
Description: The accuracy of the distal femoral varus-valgus angle was assessed by comparing the angle measured on an X-ray 12 weeks post operatively to the angle that the surgeon was targeting or planning intra operatively. A smaller number represents improved accuracy and a better outcome.
Time Frame: 12 weeks
Population: Per Protocol
Measure: Least Squares Mean (Standard Deviation); unit: Degrees
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 74 | 85
Degrees | 1.4 (1.16) | 2.0 (1.49)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; Test type: Superiority; p = 0.0058, t-test, 2 sided

3. Secondary Outcome: Accuracy of the Proximal Tibial Varus-valgus Angle Measured on Long-leg X-rays at 12 Weeks
Description: The accuracy of the proximal tibial varus-valgus angle was assessed by comparing the angle measured on an X-ray 12 weeks post operatively to the angle that the surgeon was targeting or planning intra operatively. A smaller number represents improved accuracy and a better outcome.
Time Frame: 12 weeks
Population: Per Protocol
Measure: Least Squares Mean (Standard Deviation); unit: Degrees
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 80 | 91
Degrees | 1.2 (0.95) | 1.6 (1.15)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; Test type: Superiority; p = 0.0282, t-test, 2 sided

4. Secondary Outcome: Accuracy of Femoral Component Flexion Angle Measured on Lateral X-rays at 12 Weeks
Description: The accuracy of the femoral component flexion angle was assessed by comparing the angle measured on a lateral X-ray 12 weeks post operatively to the angle that the surgeon was targeting or planning intra operatively. A smaller number represents improved accuracy and a better outcome.
Time Frame: 12 weeks
Population: Per Protocol
Measure: Least Squares Mean (Standard Deviation); unit: Degrees
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 80 | 91
Degrees | 1.9 (1.42) | 2.8 (1.89)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; Test type: Superiority; p = 0.0004, t-test, 2 sided

5. Secondary Outcome: Accuracy of the Tibial Slope Angle Measured on Lateral X-rays at 12 Weeks
Description: The accuracy of the Tibial slope angle was assessed by comparing the angle measured on a lateral X-ray 12 weeks post operatively to the angle that the surgeon was targeting or planning intra operatively. A smaller number represents improved accuracy and a better outcome.
Time Frame: 12 weeks
Population: Per Protocol
Measure: Least Squares Mean (Standard Deviation); unit: Degrees
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 80 | 91
Degrees | 1.6 (1.25) | 2.7 (2.05)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; Test type: Superiority; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Type and Frequency of Adverse Events
Description: Rate of local Adverse events and local serious adverse events reported within the first 90 days and the first year post surgery. Local means at the site of the procedure (i.e. the operated Knee). Serious adverse events are events that required medical or surgical intervention to prevent a serious impairment to health.
Time Frame: 12 weeks, 1 year
Population: Safety Analysis Set
Measure: Number; unit: Number of subjects
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 100 | 100
Number of subjects
  Number of subjects who experienced a Local Adverse Events with 1 year of the procedure. | 25 | 29
  Number of subjects who experienced a Serious Local Adverse Events within 1 year of the procedure | 6 | 16
  Number of subjects who experienced a Local Adverse Events within 90 days of the procedure | 21 | 27
  Number of subjects who experienced a Serious Local Adverse Events within 90 days of the procedure | 5 | 12
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; Comparison between the proportion of Robotic and Manual subjects who had a local adverse event within 1 year of the procedure; Test type: Superiority; p = 0.6330, Chi-squared
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; Comparison between the proportion of Robotic and Manual subjects who had a serious local adverse event within 1 year of the procedure; Test type: Superiority; p = 0.0400, Fisher Exact
Statistical Analysis 3: Comparison: Study Arm vs Control Arm; Comparison between the proportion of Robotic and Manual subjects who had a local adverse event within 90 days of the procedure; Test type: Superiority; p = 0.4079, Chi-squared
Statistical Analysis 4: Comparison: Study Arm vs Control Arm; Comparison between the proportion of Robotic and Manual subjects who had a local serious adverse event within 90 days of the procedure; Test type: Superiority; p = 0.1262, Chi-squared

7. Secondary Outcome: Soft Tissue Damage
Description: Investigators conducted an intra-operative assessment of the condition and function of key soft tissue structures in both Manual and Robotic-assisted cohorts.
Time Frame: Day of operation (intraoperative)
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 100 | 100
participants
  Incidence of medial collateral ligament being compromised intraoperatively. | 0 | 2
  Incidence of lateral collateral ligament being compromised intraoperatively. | 0 | 0
  Incidence of posterior cruciate ligament being compromised intraoperatively: number analyzed (Participants) | 62 | 28
  Incidence of posterior cruciate ligament being compromised intraoperatively | 0 | 1
  Incidence of posterior lateral capsule being compromised intraoperatively. | 0 | 0
  Incidence of posterior medial capsule being compromised intraoperatively. | 0 | 0
  Incidence of patella tendon being compromised intraoperatively. | 0 | 0

8. Other Pre Specified Outcome: EuroQol 5-Dimension 5-Level (EQ-5D-5L) - Change From Baseline
Description: The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. Scores are derived by a 5 digit code. The higher the number, the better the overall health status of the patient with 1 (meaning full health) and 0 (meaning a state as bad as being dead).
Time Frame: 1 year
Population: Per Protocol Analysis Set
  The number analyzed at each time point and for each metrics varies due to patients either being lost to follow up between visits or there being missing data during the PROM collection.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  Change from Baseline Pre op to 1 year | 0.19 (0.159) | 0.20 (0.195)
  Change from Baseline Pre op to 12 weeks: number analyzed (Participants) | 81 | 92
  Change from Baseline Pre op to 12 weeks | 0.15 (0.170) | 0.16 (0.186)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 1 year; Test type: Superiority; p = 0.6662, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 12 weeks; Test type: Superiority; p = 0.8154, t-test, 2 sided

9. Other Pre Specified Outcome: Forgotten Joint Score (FJS-12)
Description: The Forgotten Joint Scores comprise measures for the assessment of joint-specific patient-reported outcome (PRO). These PRO questionnaires focus on patients' awareness of a specific joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint. This may include strong sensations like pain, but also includes more subtle feelings like mild stiffness, subjective dysfunction, or any discomfort. The FJS-12 score ranges from 0 to 100, with 0 being the worst score and 100 being the best. A higher score means the patient is better able to forget about the artificial joint in daily life. So, the higher the score, the better the outcome is.
Time Frame: 12 weeks and 1 year
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  FJS at 12 Weeks | 35.4 (25.73) | 26.4 (23.39)
  FJS at 1 year: number analyzed (Participants) | 78 | 77
  FJS at 1 year | 53.1 (28.72) | 45.5 (33.59)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; Comparison of FJS at 12 weeks; Test type: Superiority; p = 0.0165, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; Comparison of FJS at 1 year; Test type: Superiority; p = 0.1331, t-test, 2 sided

10. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) ADL - Change From Baseline
Description: A knee-specific instrument that derives a score developed to assess the patients' opinion about their knee and associated problems. The maximum total score is 100 indicating no symptoms and the minimum is 0 indicating extreme symptoms.
Time Frame: 12 weeks, 1 year
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  Change from baseline at 1 year: number analyzed (Participants) | 78 | 75
  Change from baseline at 1 year | 35.9 (18.93) | 31.0 (23.21)
  Change from baseline at 12 weeks: number analyzed (Participants) | 86 | 92
  Change from baseline at 12 weeks | 25.6 (21.03) | 24.3 (20.07)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 1 year; Test type: Superiority; p = 0.1596, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 12 weeks; Test type: Superiority; p = 0.6834, t-test, 2 sided

11. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain - Change From Baseline
Description: as for outcome 10
Time Frame: 12 weeks, 1 year
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  Change from baseline at 1 year: number analyzed (Participants) | 78 | 76
  Change from baseline at 1 year | 37.5 (21.68) | 35.3 (24.21)
  Change from baseline at 12 weeks | 24.9 (21.91) | 25.2 (23.14)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 1 year; Test type: Superiority; p = 0.5675, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 12 weeks; Test type: Superiority; p = 0.9240, t-test, 2 sided

12. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Symptoms - Change From Baseline
Description: as for outcome 10
Time Frame: 12 weeks, 1 year
Population: Per Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  Change from baseline at 1 year | 31.1 (21.13) | 28.4 (24.02)
  Change from baseline at 12 weeks | 20.4 (21.92) | 21.8 (23.62)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 1 year; Test type: Superiority; p = 0.4586, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 12 weeks; Test type: Superiority; p = 0.6951, t-test, 2 sided

13. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Sports and Recreation - Change From Baseline
Description: as for outcome 10
Time Frame: 12 weeks, 1 year
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  Change from Baseline at 1 year: number analyzed (Participants) | 72 | 72
  Change from Baseline at 1 year | 39.5 (30.12) | 38.1 (35.09)
  Change from Baseline at 12 weeks | 23.7 (40.87) | 23.9 (30.71)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 1 year; Test type: Superiority; p = 0.8000, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 12 weeks; Test type: Superiority; p = 0.9730, t-test, 2 sided

14. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life - Change From Baseline
Description: as for outcome 10
Time Frame: 12 weeks, 1 year
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  Change from Baseline at 1 year: number analyzed (Participants) | 78 | 75
  Change from Baseline at 1 year | 45.6 (23.67) | 42.3 (31.42)
  Change from Baseline at 12 weeks | 33.4 (24.35) | 32.5 (26.28)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 1 year; Test type: Superiority; p = 0.4636, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL at 12 weeks; Test type: Superiority; p = 0.8088, t-test, 2 sided

15. Other Pre Specified Outcome: Subject Satisfaction With Knee Replacement
Description: A single patient reported question that asks the patient to score their level of satisfaction with their knee from 0-10, with 0 being fully satisfied and 10 being fully unsatisfied
Time Frame: 12 weeks, 1 year
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  Satisfaction at 12 weeks | 1.3 (2.03) | 1.6 (2.29)
  Satisfaction at 1 year: number analyzed (Participants) | 78 | 77
  Satisfaction at 1 year | 1.6 (2.73) | 1.4 (2.73)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; T-Test P-value tests the significance of the difference between ROBOTIC and MANUAL at 12 weeks; Test type: Superiority; p = 0.4851, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; T-Test P-value tests the significance of the difference between ROBOTIC and MANUAL at 1 year; Test type: Superiority; p = 0.6486, t-test, 2 sided

16. Other Pre Specified Outcome: Pain - Change From Baseline
Description: Subjects are asked how much knee pain they have had in the last week while resting (0-10) and during activity (0-10) with 0 being no pain and 10 being worst pain, therefore lower score is a better outcome.
Time Frame: 12 weeks, 1 year
Population: Per Protocol Analysis Set.
  The number analyzed at each time point and for each metrics varies due to patients either being lost to follow up between visits or there being missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 86 | 94
scores on a scale
  Pain at Rest Change from baseline at 1 year: number analyzed (Participants) | 78 | 75
  Pain at Rest Change from baseline at 1 year | -4.1 (2.93) | -4.0 (2.71)
  Pain at Rest change from baseline at 12 weeks: number analyzed (Participants) | 81 | 91
  Pain at Rest change from baseline at 12 weeks | -3.3 (3.18) | -2.9 (3.05)
  Pain at rest at 12 weeks: number analyzed (Participants) | 81 | 94
  Pain at rest at 12 weeks | 2.3 (2.38) | 3.4 (2.75)
  Pain at rest at 1 year: number analyzed (Participants) | 78 | 77
  Pain at rest at 1 year | 1.4 (2.14) | 2.1 (2.52)
  Pain with activity change from baseline at 1 year: number analyzed (Participants) | 78 | 75
  Pain with activity change from baseline at 1 year | -5.2 (2.78) | -5.0 (2.71)
  Pain with activity change from baseline at 12 weeks: number analyzed (Participants) | 81 | 91
  Pain with activity change from baseline at 12 weeks | -4.3 (2.75) | -4.0 (3.00)
  Pain with activity at 12 weeks: number analyzed (Participants) | 81 | 94
  Pain with activity at 12 weeks | 2.9 (2.43) | 3.6 (2.81)
  Pain with activity at 1 year: number analyzed (Participants) | 78 | 77
  Pain with activity at 1 year | 1.9 (2.37) | 2.5 (2.58)
Statistical Analysis 1: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline for Pain at rest between ROBOTIC and MANUAL at 1 year; Test type: Superiority; p = 0.8887, t-test, 2 sided
Statistical Analysis 2: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline for pain at rest between ROBOTIC and MANUAL at 12 weeks; Test type: Superiority; p = 0.4007, t-test, 2 sided
Statistical Analysis 3: Comparison: Study Arm vs Control Arm; T-Test P-value tests the significance of the difference between ROBOTIC and MANUAL for pain at rest at 12 weeks; Test type: Superiority; p = 0.0074, t-test, 2 sided
Statistical Analysis 4: Comparison: Study Arm vs Control Arm; T-Test P-value tests the significance of the difference between ROBOTIC and MANUAL for Pain at rest at 1 year; Test type: Superiority; p = 0.0663, t-test, 2 sided
Statistical Analysis 5: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL for Pain with Activity at 1 year; Test type: Superiority; p = 0.7096, t-test, 2 sided
Statistical Analysis 6: Comparison: Study Arm vs Control Arm; T-test P-value for difference in change from baseline between ROBOTIC and MANUAL for pain with activity at 12 weeks; Test type: Superiority; p = 0.5321, t-test, 2 sided
Statistical Analysis 7: Comparison: Study Arm vs Control Arm; T-Test P-value tests the significance of the difference between ROBOTIC and MANUAL for Pain with activity at 12 weeks; Test type: Superiority; p = 0.0709, t-test, 2 sided
Statistical Analysis 8: Comparison: Study Arm vs Control Arm; T-Test P-value tests the significance of the difference between ROBOTIC and MANUAL for Pain with activity at 1 year; Test type: Superiority; p = 0.1274, t-test, 2 sided

17. Other Pre Specified Outcome: Learning Curve
Description: The effect of learning curve on the accuracy was assessed by comparing the accuracy between the first 10 cases each surgeon completed and the subsequent cases. The accuracy was assessed by measuring the Hip-Knee-Ankle angle (HKA) on long-leg X-rays taken at 12 weeks and comparing to the planned HKA. A smaller number represents improved accuracy and a better outcome.
Time Frame: 12 Weeks
Population: Per Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Study Arm - First 10 Cases for Each Surgeon: Robotic-Assisted first 10 cases for each surgeon
- Study Arm - Latter Subjects: Robotic-Assisted cases that were performed after the first 10 for each surgeon. i.e. after the initial learning phase.
Arm/Group | Study Arm - First 10 Cases for Each Surgeon | Study Arm - Latter Subjects
Number analyzed (Participants) | 41 | 44
Degrees | 2.2 (1.66) | 2.4 (1.90)
Statistical Analysis 1: Comparison: Study Arm - First 10 Cases for Each Surgeon vs Study Arm - Latter Subjects; Comparison between the accuracy achieved in the first 10 cases compared to the subsequent cases; Test type: Superiority; p = 0.6745, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From baseline (Day 0 - including the procedure) up to the end of the study (1 year)
Description: The safety population set consisted of all enrolled participants who signed the informed consent document and attempted treatment according to the actual treatment received.
Arm/Group | Study Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 1/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 16/100 | 28/100
Other Adverse Events (participants affected / at risk) | 32/100 | 35/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=100) | Control Arm (N=100)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (9) — Local/Operative Site Events
Infection (Infections and infestations) | 0 (0) | 2 (4) — Local/Operative Site Events
Post Procedural Infection (Infections and infestations) | 0 (0) | 2 (3) — Local/Operative Site Events
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1) — Local/Operative Site Events
Bursitis Infective (Infections and infestations) | 0 (0) | 1 (1) — Local/Operative Site Events
Arthropathy disruption (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Local/Operative Site Events
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Local/Operative Site Events
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7) — Systematic - of contralateral side
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Local/Operative Site Event
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Febrileneutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Systemic Mycosis (Infections and infestations) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — On contralateral side
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonaryembolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ligament Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=100) | Control Arm (N=100)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 1 (1) | 1 (1)
Swelling (General disorders) | 0 (0) | 3 (3)
Arthritis Infection (Infections and infestations) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Use Error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 6 (6)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Noise (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 2 (2)
Device Loosening (Product Issues) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ligament Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Adverse events were coded as reported by sites per MeDRA. This resulted in some spreading of AEs. For example, "swelling" and "knee swelling" were coded differently according to best practice. Future publications will consolidate similar coded events and clarify which were combined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT04730271/Prot_SAP_003.pdf